CLINICAL TRIAL: NCT02700932
Title: Clinical Study to Evaluate the Performance of the PicoWayTM 1064 nm/ 785 nm/ 532nm Picosecond Laser for Tattoo Removal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHF20901
Record Dates: First submitted 2016-02-23; First posted 2016-03-07 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Tattoo; Pigmentation
Keywords: non-invasive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PicoWay laser treatment (Experimental): 3 wavelength tattoo treatment with picosecond laser (PicoWay)
  Interventions: Device: PicoWay

INTERVENTIONS:
Device: PicoWay — solid state laser capable of delivering energy at wavelengths of 1064 nm or 532 nm or wave length of 785±20 nm that was added to the system
  Other Names: PicoWayTM device

SUMMARY:
This is an open-label, multi-center study. Subjects in this study will receive up to eight (8) treatments in 11±5 weeks (6-16 weeks) interval, with the PicoWayTM device using the 1064 nm/ 785±20 nm/ 532 nm handpiece according to the study protocol (tattoo colors). Subjects will return for one follow-up (FU) visit at the clinic at 8 weeks following the last treatment.

Methodology described in the protocol to evaluate efficacy and safety of treatments will be carried out at each visit at the clinic

DETAILED DESCRIPTION:
This study is a prospective clinical study to demonstrate the safety and efficacy of the PicoWayTM device for tattoo removal.

Up to a total of 60 healthy candidates who are seeking tattoo removal clearance treatment from participating investigators will be enrolled at up to 3 participating study sites. Subjects will receive up to eight (8) PicoWayTM treatments at 11±5 (6-16) week's intervals. Prior to each consecutive treatment, the investigator will decide, based on degree of clearance assessment, should the subject undergo additional treatment or to be forwarded to the 8 weeks Follow-Up visit with no more treatments. Topical anesthetic (ointment) or intradermal injected solution may be used prior to treatment.

Each subject will be followed at one post treatment visit that will be conducted at:

• Eight weeks post last treatment - 8wk FU.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female and male subjects between 18 to 70 years of age
2. Fitzpatrick skin type I-VI
3. Have unwanted decorative (non-cosmetic) tattoo(s) and willing to undergo laser treatments to remove them
4. Have at least one of the following colors in the tattoo: black, green and\ or blue.
5. Willing to receive the proposed PicoWayTM treatments and comply with all study (protocol) requirements
6. Willing to have photographs and images taken of the treated areas to be used in evaluations, publications and presentations (subject identity will be masked)
7. For female subjects: not pregnant or lactating and is either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence)
8. Informed consent process is completed and subject consent is signed

Exclusion Criteria:

1. Pregnant or planning to become pregnant, having given birth less than 3 months ago, and/or breast feeding
2. Hypersensitivity to light exposure
3. Active sun tan
4. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions, hidradenitis, or dermatitis of the treatment area prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course
5. Have a history of squamous cell carcinoma or melanoma
6. History of keloid scarring, abnormal wound healing and / or prone to bruising
7. Use of oral isotretinoin (Accutane®) within 12 months of initial treatment or plans on using during the course of the study. Note: Skin must regain its normal degree of moisture prior to treatment, e.g., lack of noticeable skin flaking, skin peeling and skin surface roughness.
8. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications
9. Known allergy to lidocaine, tetracaine, Xylocaine or epinephrine
10. As per the investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Global percentage of tattoo clearance | 8 weeks post final treatment
  Global percentage of tattoo clearance as assessed by blinded evaluators based on comparing pre and post treatment photos.

SECONDARY OUTCOMES:
Rate of tattoo clearance | 8 weeks post final treatment
  Average number of treatments determined to achieve 50 and 75 percent clearance
Adverse event reporting | Through study completion, average of 1 year
  Based on rate and severity of treatments with the PicoWay laser treatment

CONTACTS AND LOCATIONS:
Overall Officials: Eric F Bernstein, MD, Principal Investigator — Main Line Center for Laser Surgery
Locations (1):
- Main Line Center for Laser Surgery, Ardmore, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bernstein EF, Schomacker KT, Basilavecchio LD, Plugis JM, Bhawalkar JD. A novel dual-wavelength, Nd:YAG, picosecond-domain laser safely and effectively removes multicolor tattoos. Lasers Surg Med. 2015 Sep;47(7):542-548. doi: 10.1002/lsm.22391. Epub 2015 Jul 14. PMID 26175187
- [Background] Saedi N, Metelitsa A, Petrell K, Arndt KA, Dover JS. Treatment of tattoos with a picosecond alexandrite laser: a prospective trial. Arch Dermatol. 2012 Dec;148(12):1360-3. doi: 10.1001/archdermatol.2012.2894. PMID 22986470